CLINICAL TRIAL: NCT05127954
Title: A Multicenter, Open-label, Extension Study to Evaluate the Long-term Safety and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine With or Without Aura in Children and Adolescents (Ages 6-17)
Brief Title: Long-term Extension Study to Assess Safety and Tolerability of Oral Ubrogepant Tablets for the Acute Treatment of Migraine in Pediatric Participants (Ages 6-17)
Acronym: UBRO PEDS OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3110-306-002
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: Migraine; Ubrogepant; Ubrelvy
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ubrogepant Dose A (12 to 17 Years Old) (Experimental): Participants will receive oral tablets of ubrogepant Dose A for qualifying migraine attack. Participants have the option to take a second dose of ubrogepant or rescue medication, at least 2 hours after initial dose for headache of any intensity.
  Interventions: Drug: Ubrogepant
- Ubrogepant Dose B (6 to 11 Years Old) (Experimental): Participants will receive the highest dose of oral tablets of ubrogepant tested in Study 3110-305-002 for qualifying migraine attack. Participants have the option to take a second dose of ubrogepant or rescue medication, at least 2 hours after initial dose for headache of any intensity.
  Interventions: Drug: Ubrogepant

INTERVENTIONS:
Drug: Ubrogepant — Oral Tablet
  Other Names: Ubrelvy

SUMMARY:
Migraine is a common neurological disorder typically characterized by attacks of throbbing, moderate to severe headache, often associated with nausea, vomiting, and sensitivity to light and sound. Migraine is extremely common and disabling in children. The purpose of this study is to evaluate long term safety and tolerability of ubrogepant in the acute treatment of migraine in pediatric participants.

Ubrogepant is a drug approved for the acute treatment of migraine in adults. Pediatric participants (aged 6-17 years) with a history of migraine will be enrolled. Participants who completed the lead-in Study 3110-305-002, as well as those who were placebo responders and screen failed, will be eligible to enroll into this study. Around 1200 participants will be enrolled in the study at approximately 120 sites in the United States.

Participants may receive ubrogepant oral tables to treat up to 8 migraine attacks of any intensity per month. There will be an option to take a second dose of study intervention (identical to initial dose), or rescue medication, starting 2 hours after the initial dose. The study duration will be up to 54 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The safety and tolerability of the treatment will be checked by medical assessments, blood tests, checking for adverse events and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Completers of the lead-in Study 3110-305-002 (in the main study or PK cohort) or those who screen failed due to being placebo responders.
* Demonstrated an acceptable degree of compliance with study procedures in the lead-in study and who, in the investigator's clinical judgment, did not experience an AE that may indicate an unacceptable safety risk for this study.

Exclusion Criteria:

* Requirement for any medication (eg, barbiturates) or diet (eg, grapefruit juice) that is on the list of prohibited concomitant medications that cannot be discontinued or switched to an allowable, alternative medication at Visit 1.
* An ECG with clinically significant abnormalities at Visit 1 as determined by the investigator.
* Clinically significant abnormalities in physical examination at Visit 1, as determined by the investigator.
* Significant risk of self-harm, based on clinical interview and responses on the C-SSRS, or of harm to others in the opinion of the investigator; participants should be excluded if they report suicidal ideation with intent, with or without a plan (ie, Type 4 or 5 on the C-SSRS), or report suicidal behavior at Visit 1
* Any medical or other reason (eg, unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study) that, in the investigator's opinion, might indicate that the participant is unsuitable for the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | up to 54 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants with Potentially Clinically Significant Clinical 12-lead Electrocardiogram (ECG) | Up to 54 Weeks
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Percentage of Participants with Potentially Clinically Significant Vital Sign Parameters | Up to 54 Weeks
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Percentage of Participants with Potentially Clinically Significant lab values | Up to 54 Weeks
  Percentage of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Percentage of with Participants with Suicidal Ideation or Suicidal Behavior | Up to 54 Weeks
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation was classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt).
Percentage of Participants with Change in Menstrual Cycle | Up to 54 Weeks
  Female participants who have entered menarche are to be asked for the date of the first and last day of their most recent menstrual period.
Change from baseline in Tanner staging score | Up to 54 Weeks
  Tanner's staging is used to assess growth and pubertal development.
Change From baseline in Behavior Rating Inventory of Executive Function (BRIEF 2) questionnaire | up to 54 weeks
  The BRIEF 2 is an 86-item questionnaire assessing executive function. It consists of 2 indexes, Behavioral Regulation and Metacognition, which are then used to calculate an overall composite score. Higher scores indicate more executive difficulties

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (113):
- United States (109):
  - Rehabilitation & Neurological Services /ID# 240054, Huntsville, Alabama
  - The Center for Clinical Trials - Saraland /ID# 239448, Saraland, Alabama
  - Preferred Research Partners /ID# 238979, Little Rock, Arkansas
  - Advanced Research Center /ID# 238967, Anaheim, California
  - Neuro Pain Medical Center /ID# 239135, Fresno, California
  - Alliance for Research Alliance for Wellness /ID# 233497, Long Beach, California
  - Children's Hospital Los Angeles /ID# 239446, Los Angeles, California
  - Excell Research, Inc /ID# 233495, Oceanside, California
  - Paradigm Clinical Research - San Diego /ID# 269611, San Diego, California
  - Lumos Clinical Research Center /ID# 239018, San Jose, California
  - Pacific Clinical Research Management Group /ID# 238503, Upland, California
  - Sunwise Clinical Research /ID# 238458, Walnut Creek, California
  - Children's Hospital Colorado - Aurora /ID# 239838, Aurora, Colorado
  - IMMUNOe Research Centers /ID# 240846, Centennial, Colorado
  - MCB Clinical Research Centers /ID# 240999, Colorado Springs, Colorado
  - New England Institute for Clinical Research /ID# 239019, Stamford, Connecticut
  - Emerson Clinical Research Inst /ID# 238455, Washington D.C., District of Columbia
  - Encore Medical Research of Boynton Beach LLC /ID# 248720, Boynton Beach, Florida
  - Gulf Coast Clinical Research Center /ID# 233335, Fort Myers, Florida
  - Sarkis Clinical Trials /ID# 233493, Gainesville, Florida
  - Northwest Florida Clinical Research Group, LLC /ID# 244396, Gulf Breeze, Florida
  - A.G.A Clinical Trials /ID# 238409, Hialeah, Florida
  - Encore Medical Research /ID# 247463, Hollywood, Florida
  - Advanced Research Institute of Miami /ID# 240712, Homestead, Florida
  - Auzmer Research /ID# 241514, Lakeland, Florida
  - Columbus Clinical Services, Llc /Id# 238968, Miami, Florida
  - My Preferred Research LLC /ID# 239020, Miami, Florida
  - Neurology & Pain Medicine /ID# 241860, Miami, Florida
  - Medical Research Group of Central Florida /ID# 240711, Orange City, Florida
  - Clinical Associates of Orlando, LLC /ID# 272623, Orlando, Florida
  - Suncoast Clinical Research - Palm Harbor /ID# 233535, Palm Harbor, Florida
  - Asclepes Research Centers - Spring Hill /ID# 231872, Spring Hill, Florida
  - University of South Florida- Neuroscience Institute /ID# 233420, Tampa, Florida
  - Encore Medical Research - Weston /ID# 248335, Weston, Florida
  - Pediatric Neurology and Epilepsy Specialists /ID# 233336, Winter Park, Florida
  - Global Research Associates /ID# 243504, Atlanta, Georgia
  - Rare Disease Research, LLC /ID# 238833, Atlanta, Georgia
  - Clinical Integrative Research Center of Atlanta (CIRCA) /ID# 238852, Atlanta, Georgia
  - Coastal Georgia Child Neurology /ID# 240845, Brunswick, Georgia
  - CenExcel iResearch LLC /ID# 239832, Decatur, Georgia
  - Velocity Clinical Research - Savannah /ID# 231873, Savannah, Georgia
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 238454, Stockbridge, Georgia
  - Velocity Clinical Research - Boise /ID# 238978, Meridian, Idaho
  - Chicago Headache Center & Research Institute /ID# 254071, Chicago, Illinois
  - Accellacare - McFarland Clinic /ID# 238490, Ames, Iowa
  - College Park Family Care Center Overland Park /ID# 240707, Overland Park, Kansas
  - Clinical Associates Midwest, LLC /ID# 274356, Overland Park, Kansas
  - Psychiatric Associates /ID# 240710, Overland Park, Kansas
  - Alliance for Multispecialty Research (AMR) - Wichita West /ID# 239829, Wichita, Kansas
  - University of Kentucky Chandler Medical Center /ID# 233428, Lexington, Kentucky
  - Pharmasite Research, Inc. /ID# 233414, Baltimore, Maryland
  - Minneapolis Clinic of Neurology - Burnsville /ID# 238828, Burnsville, Minnesota
  - MediSync Clinical Research Hattiesburg Clinic /ID# 239837, Petal, Mississippi
  - Proven Endpoints LLC /ID# 240974, Ridgeland, Mississippi
  - Sharlin Health Neuroscience Research Center /ID# 238969, Ozark, Missouri
  - Cognitive Clinical Trials (CCT) - Papillion /ID# 239835, Papillion, Nebraska
  - Healthy Perspectives - Innovative Mental Health Services, PLLC /ID# 239441, Nashua, New Hampshire
  - Hunterdon Neurology /ID# 248222, Annandale, New Jersey
  - Goryeb Children's Hospital /ID# 239425, Morristown, New Jersey
  - CVS HealthHUB - Runnemede /ID# 240057, Runnemede, New Jersey
  - Dent Neurologic Institute - Amherst /ID# 238415, Amherst, New York
  - Bioscience Research /ID# 239442, Mount Kisco, New York
  - Modern Migraine MD /ID# 263140, New York, New York
  - North Suffolk Neurology /ID# 238457, Port Jefferson Station, New York
  - SUNY Upstate Medical University /ID# 241140, Syracuse, New York
  - CVS HealthHUB - Charlotte /ID# 240842, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC - Hickory /ID# 238946, Hickory, North Carolina
  - Patient Priority Clinical Sites, LLC /ID# 240051, Cincinnati, Ohio
  - University of Cincinnati /ID# 238461, Cincinnati, Ohio
  - Cincinnati Childrens Hospital Medical Center /ID# 247491, Cincinnati, Ohio
  - Headache Center of Hope /ID# 244819, Cincinnati, Ohio
  - Centricity Research Columbus /ID# 238832, Columbus, Ohio
  - CincyScience /ID# 233334, West Chester, Ohio
  - IPS Research Company /ID# 231876, Oklahoma City, Oklahoma
  - Providence Brain and Spine Institute /ID# 240050, Portland, Oregon
  - Children's Hospital of Philadelphia - Main /ID# 241138, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC - Scottdale /ID# 239017, Scottdale, Pennsylvania
  - Frontier Clinical Research - Smithfield /ID# 238502, Smithfield, Pennsylvania
  - Coastal Pediatric Research /ID# 240708, Charleston, South Carolina
  - Tribe Clinical Research LLC /ID# 239143, Greenville, South Carolina
  - Duplicate_Premier Neurology, P.C. /ID# 233419, Greer, South Carolina
  - Access Clinical Trials, Inc. /ID# 238414, Nashville, Tennessee
  - UT Health Austin at Dell Children's Neurology Clinic /ID# 246570, Austin, Texas
  - BioBehavioral Research of Austin /ID# 233427, Austin, Texas
  - Velocity Clinical Research, Austin /ID# 233406, Austin, Texas
  - Tekton Research - Beaumont /ID# 238407, Beaumont, Texas
  - Relaro Medical Trials /ID# 241141, Dallas, Texas
  - Cedar Health Research /ID# 233403, Dallas, Texas
  - 3A Research - East El Paso /ID# 241665, El Paso, Texas
  - Earle Research /ID# 238940, Friendswood, Texas
  - DM Clinical Research /ID# 238361, Houston, Texas
  - Houston Clinical Research Associates /ID# 246522, Houston, Texas
  - Sante Clinical Research /ID# 248333, Kerrville, Texas
  - FMC Science /ID# 240475, Lampasas, Texas
  - Livingspring Family Medical Center /ID# 252194, Mansfield, Texas
  - AIM Trials /ID# 233425, Plano, Texas
  - Road Runner Research /ID# 238360, San Antonio, Texas
  - Family Psychiatry of The Woodlands /ID# 238980, The Woodlands, Texas
  - ClinPoint Trials /ID# 238406, Waxahachie, Texas
  - Pantheon Clinical Research /ID# 251475, Bountiful, Utah
  - Highland Clinical Research /ID# 240053, Salt Lake City, Utah
  - University of Utah Health Hospital /ID# 239021, Salt Lake City, Utah
  - Neuropsychiatric Associates LLC/DBA Woodstock Research Center /ID# 240055, Woodstock, Vermont
  - Office of Maria Ona /ID# 239833, Franklin, Virginia
  - Children's Hospital of The King's Daughters - Children's Medical Tower /ID# 239142, Norfolk, Virginia
  - National Clinical Research /ID# 238419, Richmond, Virginia
  - Core Clinical Research /ID# 233421, Everett, Washington
  - Frontier Clinical Research - Kingwood /ID# 238459, Kingwood, West Virginia
  - Mind+ Neurology /ID# 275538, Mequon, Wisconsin
- Puerto Rico (4):
  - Clinical Research Investigator Group, LLC /ID# 267458, Bayamón
  - Puerto Rico Health Institute /ID# 250560, Dorado
  - GCM Medical Group PSC /ID# 250561, San Juan
  - Caribbean Medical Research Center /ID# 265292, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/